CLINICAL TRIAL: NCT03058718
Title: Effectiveness of Procalcitonin-Guided Antibiotic Therapy in Acute Exacerbations of Bronchiectasis: a Randomized Controlled Trial
Brief Title: Procalcitonin-Guided Antibiotic Therapy in Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Qian Qi, assistant director, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: lwsrmyy
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Procalcitonin; Bronchiectasis; Antibiotic Therapy
MeSH Terms: conditions — Bronchiectasis | interventions — Procalcitonin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Procalcitonin-guided antibiotic treatment group (Experimental): Patients were divided into 2 subgroups:
  1. No infection group (including patients with procalcitonin<0.1 ng/ml at enrollment, and patients with 0.1 ng/ml ≤procalcitonin ≤0.25 ng/ml at enrollment who are with stable respiratory and hemodynamics, and without serious complications) : the group is not given the application of antibiotics.
  2. Infection group (including patients with procalcitonin>0.25 ng/ml at the time of enrollment, and patients with 0.1 ng/ml ≤ procalcitonin≤0.25 ng/ml at enrollment who have severe disease, unstable hemodynamics, and severe complications or intensive care unit treatment): the group is given the application of antibiotics. According to the guidelines for severe sepsis / septic shock treatment, the standard for discontinuation of antimicrobial agents: If the procalcitonin level falls below <0.1 ng/ml or more than 80%, compared with the baseline before enrollment, it is recommended to discontinue the antimicrobial agent.
  Interventions: Other: Procalcitonin
- Standard antibiotic therapy group (Active Comparator): The application of antibiotics is given to patiens according to the doctor's experience.
  Interventions: Other: Clinical Experience

INTERVENTIONS:
Other: Procalcitonin — The application of antimicrobial agents is determined by PCT results.
  Arms: Procalcitonin-guided antibiotic treatment group
Other: Clinical Experience — The application of antimicrobial agents is determined by clinical experience of doctors.
  Arms: Standard antibiotic therapy group

SUMMARY:
To explore effectiveness of procalcitonin-guided antibiotic therapy in acute exacerbations of bronchiectasis, and to explore the clinical value of procalcitonin in bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

1. Bronchiectasis was diagnosed by high-resolution computed tomography based on the criteria published by McShane PJ et al.
2. Acute exacerbations of bronchiectasis.
3. Aged >= 18 years.
4. Procalcitonin been detected after admission.

Exclusion Criteria:

1. Associated with chronic obstructive pulmonary disease.
2. Associated with asthma.
3. Traction bronchiectasis caused by pulmonary fibrosis.
4. Rule out other possible cause procalcitonin increased diseases such as cancer, connective tissue disease, active tuberculosis, chronic liver disease and respiratory system than the bacterial infection.
5. Clinical data were incomplete.
6. Can not follow up with the person.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Antimicrobial prescription rate | 14 days
Number of days of antimicrobial application | 14 days
The number of days in hospital | 14 days

SECONDARY OUTCOMES:
Effective rate of clinical treatment | 14 days
Quality of life score | 6 months
Adverse reaction rate | 14 days
Bacterial resistance rate | 14 days
The incidence of complications | 14 days
fungal infection rate | 14 days
mortality rate | 14 days
The proportion of patients with at least once acute exacerbation in 6 months | 6 months